CLINICAL TRIAL: NCT04844021
Title: A Comparative Effectiveness Trial of Strategies to Implement Firearm Safety Promotion as a Universal Suicide Prevention Strategy in Pediatric Primary Care
Brief Title: Adolescent and Child Suicide Prevention in Routine Clinical Encounters
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Pennsylvania (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rinad Beidas, Ralph Seal Paffenbarger Professor and Chair, Department of Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH123491 (NIH); R01MH123491 (NIH)
Record Dates: First submitted 2020-11-18; First posted 2021-04-14 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Suicide
Keywords: implementation; fidelity; facilitation; firearm
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: The investigators will randomize clinics to the active implementation conditions (Nudge [k = 15] or Nudge+ [k = 15]). Clinicians in clinics assigned to both conditions will deliver the S.A.F.E. Firearm storage program to patients during well-child visits.
  Clinicians from all participating clinics, regardless of study arm, will be invited to participate in surveys and interviews.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nudge (Experimental): Clinics randomized to the Nudge condition will receive the EHR prompt only. The investigators will add default language to the standard Well Child Visit workflow to serve as a reminder and allow for tracking of S.A.F.E. Firearm implementation. The clinician will be asked to denote whether the program was delivered (e.g., whether conversation around firearm storage was conducted, whether cable firearm lock was offered) to the parent during the visit. This EHR prompt will remain turned "on" from active implementation through the sustainment period.
  Interventions: Behavioral: Nudge
- Nudge+ (Experimental): This arm consists of Nudge as described above, as well as facilitation. Facilitation (i.e., external support delivered by health system employees not employed within the clinic site) will be offered for 12 months to each clinic, in keeping with other implementation trials. The investigators will use a train-the-trainer model to train facilitators at both health systems to ensure they achieve facilitator core competencies with an eye toward implementation of S.A.F.E. Firearm. The role of the facilitator is to engage with study clinics, to assist each clinic in setting change and performance goals around the implementation of S.A.F.E. Firearm, and to troubleshoot implementation barriers.
  Interventions: Behavioral: Nudge+

INTERVENTIONS:
Behavioral: Nudge — EHR-based "nudge"
  Arms: Nudge
Behavioral: Nudge+ — EHR-based "nudge" plus facilitation
  Arms: Nudge+

SUMMARY:
The objective of this study is to compare two approaches to implement an evidence-based firearm safety promotion program, S.A.F.E. Firearm, in pediatric primary care as a universal suicide prevention strategy. The first implementation approach is a prompt in the electronic health record (EHR; Nudge) reminding clinicians to a) discuss firearm storage and b) offer a free cable firearm lock during the pediatric well visit. The second implementation approach (Nudge+) includes both the EHR Nudge described above plus one year of support to the clinics in deploying the program (i.e., practice facilitation). The study also aims to identify how these strategies work and whether the S.A.F.E. Firearm program results in reduced unauthorized access to firearms by young people. The investigators hypothesize that a greater proportion of well-visits will have S.A.F.E. Firearm delivery documented in the electronic health record in Nudge+ clinics vs. Nudge clinics.

DETAILED DESCRIPTION:
The investigators will conduct a hybrid type III effectiveness-implementation trial using a longitudinal cluster randomized design to test the most effective way to implement S.A.F.E. Firearm among 30 clinics, 158 clinicians, and 48,475 youth nested in two Mental Health Research Network (MHRN) health systems in Michigan and Colorado. Clinics will be randomized to receive either the EHR implementation strategy (Nudge) or the EHR implementation strategy plus 1 year of facilitation to target implementation barriers (Nudge+).

Aim 1: Examine the effects of Nudge vs. Nudge+ on implementation outcomes.

* Reach: The investigators hypothesize that clinician-documented program delivery in the EHR (reach; primary outcome) will be superior in the Nudge+ condition compared to Nudge in the active and sustainment periods.
* Fidelity: The investigators hypothesize that parent-reported clinician fidelity to the program will be superior in the Nudge+ condition compared to Nudge in the active and sustainment periods.
* Cost: The investigators will also assess implementation strategy cost.
* Cable Locks/Acceptability: The investigators hypothesize that the Nudge+ condition will result in increased rates of cable lock distribution and higher acceptability compared with Nudge in both the active and sustainment periods.

Aim 2: Use mixed methods to identify implementation strategy mechanisms. The investigators hypothesize that Nudge+ will have a stronger effect because it will improve clinic adaptive reserve (i.e., the ability to make and sustain change). The investigators will also investigate the role of clinician motivation. The investigators hypothesize that clinician attitudes towards firearm counseling, clinician burnout, and clinician demographics will moderate implementation strategy effectiveness.

Aim 3: Examine the effects of the adapted intervention on clinical outcomes. The investigators hypothesize that Nudge+ will result in a greater proportion of parents reporting that they made firearm(s) less accessible to their child(ren) compared with Nudge. The investigators will explore rates of youth suicide attempts, deaths, and unintentional firearm injury and mortality by implementation condition and across time.

ELIGIBILITY:
Inclusion Criteria: Parents

* Parents and/or legal guardians (hereafter referred to as parents) at participating pediatric clinics who have a child age 5-17 who attends a well visit. At least one parent must attend the well visit to be eligible. The parent must be at least 18 years old to participate.

Exclusion Criteria: Parents

* Due to translation costs and challenges of recruiting non-US resident participants, respectively, non-English speaking parents and non-US resident parents will not be eligible to participate at Henry Ford Health System.

Inclusion Criteria: Clinicians and leaders

* Pediatric physicians and non-physician clinicians (hereafter referred to as clinicians) employed within the participating pediatric clinics, as well as health system leaders employed within the two health systems, are eligible to participate. Family medicine clinicians who see pediatric patients in participating clinics at Kaiser Permanente Colorado will also be eligible.

Exclusion criteria: Clinicians and leaders

* At Kaiser Permanente Colorado, family medicine clinicians whose patient panel is comprised of fewer than 5% pediatric patients will be excluded.
* Family medicine clinicians who see pediatric patients in participating clinics at Henry Ford Health System will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47307 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kaiser Permanente Colorado, Aurora, Colorado
  - Henry Ford Health System, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Waller CR, Pandey M, Boggs JM, Beck A, Bedoy RP, Buttenheim AM, Elias ME, Hoskins K, Jager-Hyman S, Johnson C, Maye M, McArdle B, Pappas C, Small DS, Quintana LM, Wolk CB, Wright LA, Williams NJ, Ahmedani BK, Beidas RS. Pediatric Healthcare Worker Perspectives on Implementation of a Secure Firearm Storage Program: A Qualitative Study. Res Sq [Preprint]. 2025 Oct 8:rs.3.rs-7437500. doi: 10.21203/rs.3.rs-7437500/v1. PMID 41282060
- [Derived] Beidas RS, Linn KA, Boggs JM, Marcus SC, Hoskins K, Jager-Hyman S, Johnson C, Maye M, Quintana L, Wolk CB, Wright L, Pappas C, Beck A, Bedjeti K, Buttenheim AM, Daley MF, Elias M, Lyons J, Martin ML, McArdle B, Ritzwoller DP, Small DS, Williams NJ, Zhang S, Ahmedani BK. Implementation of a Secure Firearm Storage Program in Pediatric Primary Care: A Cluster Randomized Trial. JAMA Pediatr. 2024 Nov 1;178(11):1104-1113. doi: 10.1001/jamapediatrics.2024.3274. PMID 39226027
- [Derived] Beidas RS, Ahmedani BK, Linn KA, Marcus SC, Johnson C, Maye M, Westphal J, Wright L, Beck AL, Buttenheim AM, Daley MF, Davis M, Elias ME, Jager-Hyman S, Hoskins K, Lieberman A, McArdle B, Ritzwoller DP, Small DS, Wolk CB, Williams NJ, Boggs JM. Study protocol for a type III hybrid effectiveness-implementation trial of strategies to implement firearm safety promotion as a universal suicide prevention strategy in pediatric primary care. Implement Sci. 2021 Sep 22;16(1):89. doi: 10.1186/s13012-021-01154-8. PMID 34551811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We included children (ages 5-17) attending an in-person well-child visit at a participating pediatric clinic from March 14, 2022 until March 20, 2023. Demographic information and outcomes were assessed for all eligible visits during the study period (e.g., demographic information for two well-child visits with the same patient are included as two separate "participants" in our demographic descriptive statistics). Data were extracted from the electronic health record (EHR).
Pre-assignment Details: Randomization was at clinic level. Clinics and all clinicians at them received Nudge or Nudge+. Clinics and clinicians are NOT considered "enrolled participants" in our primary outcomes analysis. Parents attending visits with the child received S.A.F.E. Firearm from clinicians, but are NOT considered "enrolled participants" in our primary outcomes analysis. Units of analysis for the primary outcome are number of visits; thus, "participants" in this participant flow refers to well-child visits.
Units Other Than Participants: clinics
Groups:
- Nudge: Clinics randomized to the Nudge condition will receive the EHR prompt only. The investigators will add default language to the standard Well Child Visit workflow to serve as a reminder and allow for tracking of S.A.F.E. Firearm implementation. The clinician will be asked to denote whether the program was delivered (e.g., whether conversation around firearm storage was conducted, whether cable firearm lock was offered) to the parent during the visit.
- Nudge+: This arm consists of Nudge as described, as well as facilitation. Facilitation (i.e., external support delivered by health system employees not employed within the clinic site) will be offered for 12 months to each clinic, in keeping with other implementation trials. The role of the facilitator is to engage with study clinics, to assist each clinic in setting change and performance goals around the implementation of S.A.F.E. Firearm, and to troubleshoot implementation barriers.
Period: Overall Study
Arm/Group | Nudge | Nudge+
Started | 24989; 15 clinics | 22318; 15 clinics
Completed | 24989; 15 clinics | 22318; 14 clinics
Not Completed | 0; 0 clinics | 0; 1 clinics

BASELINE CHARACTERISTICS:
Population: "Participants" refers to well-child visits with patients ages 5-17. Data were extracted from the electronic health record (EHR).
Groups:
- Total: Total of all reporting groups
Arm/Group | Nudge | Nudge+ | Total
Number analyzed (Participants) | 24989 | 22318 | 47307
Age, Continuous [Mean (Standard Deviation); unit: years] — Patient age in years
  years | 11.122 (3.718) | 11.448 (3.703) | 11.276 (3.714)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Patient sex assigned at birth
  Participants
    Sex: female | 12143 | 10948 | 23091
    Sex: male | 12843 | 11367 | 24210
    Sex: unknown | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Patient ethnicity
  Participants
    Hispanic or Latino | 2459 | 3879 | 6338
    Not Hispanic or Latino | 19966 | 16580 | 36546
    Unknown or Not Reported | 2564 | 1859 | 4423
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Patient race: White | 10741 | 11181 | 21922
  Patient race: Black or African American | 7013 | 3438 | 10451
  Patient race: Asian | 1154 | 1348 | 2502
  Patient race: Native American or Alaska Native | 94 | 79 | 173
  Patient race: Native Hawaiian or Other Pacific Islander | 33 | 49 | 82
  Patient race: Other race | 1471 | 1210 | 2681
  Patient race: More than one race | 781 | 937 | 1718
  Patient race: Unknown | 3702 | 4076 | 7778

OUTCOME MEASURES:

1. Primary Outcome: Reach
Description: Reach is the proportion of eligible well-child visits who received the S.A.F.E. Firearm program. "Participants" refers to well-child visits. For each well-child visit, data regarding S.A.F.E. Firearm delivery were available in the form of binary indicators, with 1 indicating S.A.F.E. Firearm was delivered during the visit and 0 indicating S.A.F.E. Firearm was not delivered during the visit. Reach outcomes presented below are means of the binary indicators, which were calculated across all eligible well-child visits.
Time Frame: EHR data on reach will be extracted for the time period: the beginning of the active implementation period through the end of the active implementation period (12 months total)
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: proportion of visits
Arm/Group | Nudge | Nudge+
Number analyzed (Participants) | 24989 | 22318
proportion of visits | 0.2735 [0.2680 to 0.2790] | 0.4045 [0.3981 to 0.4109]
Statistical Analysis 1: Comparison: Nudge; The primary analysis involved fitting generalized estimating equations (GEE) with a binomial distribution and logit link to estimate reach (primary endpoint) for Nudge and Nudge+ along with the risk difference between conditions; Test type: Other — We used a multiple hypothesis testing framework to evaluate the effectiveness of Nudge+ vs. Nudge, considering: 1) Nudge+ is more effective than Nudge by over 10 percentage points (PP); 2) Nudge+ is as effective as Nudge, with a difference of no greater than 10 PP in either direction; and 3) Nudge+ is less effective than Nudge by over 10 PP. The 10 PP margin was selected based on discussions with health system leaders and previous studies to ensure the differences were clinically meaningful; If the 95% confidence interval for the risk difference did not contain any values within a region (Nudge+ superior, equivalence, Nudge+ inferior), that region could be rejected; Marginal probability = 0.22, 95% CI 2-sided [0.13 to 0.31]
Statistical Analysis 2: Comparison: Nudge+; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; [p-value comment as in outcome 1, analysis 1]; Marginal probability = 0.49, 95% CI 2-sided [0.37 to 0.61]

2. Secondary Outcome: Fidelity
Description: Whether the clinician followed the two S.A.F.E. Firearm steps (counseling and offering cable lock), measured via parent-report
Time Frame: surveys collected from parents within two weeks of well-child visit. Surveys will be collected during the duration of the pre-implementation, active implementation, and sustainment phases (30 months total)
Reporting Status: Not Posted

3. Secondary Outcome: Parent-reported Acceptability
Description: Parent-report of acceptability of the S.A.F.E. Firearm program. Parents will be asked to answer questions pertaining to the acceptability of program components. Specifically, they will answer yes/no questions developed by the research team which ask whether they found the component acceptable.
Time Frame: Parent surveys will be collected from parents within two weeks of well-child visit from pre-implementation through sustainment (30 months total)
Reporting Status: Not Posted

4. Secondary Outcome: Clinician-reported Acceptability
Description: Clinician-report of acceptability of the S.A.F.E. Firearm program. Acceptability of the implementation strategies - EHR nudge and facilitation - will be collected from clinicians as well. Clinicians will be asked questions developed by the research team about whether they found various components of the program and implementation strategies acceptable, and will answer each question with a Likert-scaled answer.
Time Frame: Clinician surveys will be collected at two time points during the study period: during pre-implementation (surveys will be administered for approximately 1 month) and during active implementation (surveys will be administered for approximately 1 month)
Reporting Status: Not Posted

5. Secondary Outcome: Cost
Description: Cost of the implementation strategies (EHR nudge, facilitation) and the S.A.F.E. Firearm program delivery. Data on the cost of implementing the program (e.g., costs for printing program materials and distributing firearm locks) and the implementation strategies (e.g., facilitator full-time equivalent [FTE] time) will be collected to estimate the overall cost of the program and implementation strategy delivery.
Time Frame: Cost data will be collected from pre-implementation through sustainment (30 months total)
Reporting Status: Not Posted

6. Secondary Outcome: Distribution of Cable Locks
Description: Number of cable locks distributed by each clinic will be collected
Time Frame: Cable lock distribution data will be collected from active implementation through sustainment (24 months total)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Description: Our enrolled participants were well-child visits; "number affected" and "number at risk" refers to well-child visits. Adverse event information is reported for all eligible well-child visits during the study period (e.g., information for two well-child visits with the same patient are included as two separate "at-risk participants" in our demographic descriptive statistics).
Arm/Group | Nudge | Nudge+
All-Cause Mortality (participants affected / at risk) | 0/24989 | 0/22318
Serious Adverse Events (participants affected / at risk) | 0/24989 | 0/22318
Other Adverse Events (participants affected / at risk) | 0/24989 | 0/22318

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT04844021/Prot_001.pdf
  • Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT04844021/SAP_002.pdf
  • Informed Consent Form (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT04844021/ICF_000.pdf